CLINICAL TRIAL: NCT01945489
Title: OnabotulinumtoxinA (BOTOX®) Treatment for Urinary Incontinence in Patients With Overactive Bladder
Acronym: COMFORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GMA-OAB-113
Record Dates: First submitted 2013-09-16; First posted 2013-09-18 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-09

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OnabotulinumtoxinA (Experimental): OnabotulinumtoxinA (BOTOX®) 100U injected into the detrusor at Day 1, followed by a repeat injection of onabotulinumtoxinA 100U after a minimum of 12 weeks (if applicable).
  Interventions: Biological: onabotulinumtoxinA
- Placebo/OnabotulinumtoxinA (Other): Placebo (Normal saline) injected into the detrusor on Day 1, followed by an injection of onabotulinumtoxinA 100U after a minimum of 12 weeks (if applicable).
  Interventions: Biological: onabotulinumtoxinA; Drug: Normal saline

INTERVENTIONS:
Biological: onabotulinumtoxinA — OnabotulinumtoxinA (BOTOX®) injected into the detrusor.
  Other Names: BOTOX®; botulinum toxin Type A
Drug: Normal saline — Normal saline (placebo) injected into the detrusor.
  Arms: Placebo/OnabotulinumtoxinA

SUMMARY:
This is a study to evaluate the efficacy and safety of onabotulinumtoxinA (BOTOX®) compared with placebo, in achieving a 100% reduction in urinary incontinence in patients with overactive bladder (OAB) not properly managed with an anticholinergic.

ELIGIBILITY:
Inclusion Criteria:

-Patients with symptoms of Overactive Bladder (OAB) (frequency and urgency) with urinary incontinence for at least 6 months prior to screening.

Exclusion Criteria:

* Symptoms of OAB due to a neurological reason
* Use of anticholinergics or other medications or therapies to treat symptoms of OAB within 7 days of screening
* Use of Clean Intermittent Catheterization (CIC) or indwelling catheter to manage urinary incontinence
* Use of botulinum toxin therapy of any serotype for any urological condition
* Use of botulinum toxin therapy of any serotype for any non-urological condition in the 12 weeks prior to screening
* History of any pelvic or urological abnormalities, bladder surgery or disease, other than OAB, that may affect bladder function
* Diagnosis of Myasthenia gravis, Eaton-Lambert syndrome, or Amyotrophic Lateral Sclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2017-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Aboushwareb, Study Director — Allergan
Locations (40):
- United States (40):
  - Urologic Clinics of North Alabama, Huntsville, Alabama
  - Alaska Urological Institute dba Alaska Clinical Research Center, Anchorage, Alaska
  - South Orange County Medical Research Center, Laguna Hills, California
  - University of Southern California, Los Angeles, California
  - Genesis Research LLC, San Diego, California
  - U. Colorado, School of Med., Aurora, Colorado
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Urology Associates of Norwalk, Norwalk, Connecticut
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - Bladder and Prostate Health Investigations, LLC, Miramar, Florida
  - Renstar Medical Research, Ocala, Florida
  - Urology Health Team, PLLC, Ocala, Florida
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Atlanta Medical Research Institute, Alpharetta, Georgia
  - Northeast Indiana, Fort Wayne, Indiana
  - Urogynecology Associates, Indianapolis, Indiana
  - Deaconess Clinic, Inc., Newburgh, Indiana
  - Urology of Indiana, LLC, Noblesville, Indiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Owings Mills, Maryland
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Accumed Research, Garden City, New York
  - Manhattan Medical Research, New York, New York
  - Premier Medical Group of the Hudson Valley, Newburgh, New York
  - Advanced Urology Centers of NY A division of IMP, Plainview, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Associated Medical Professionals of New York, PLLC, Syracuse, New York
  - Carolina Urology Partners, PLLC, Gastonia, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - TriState Urologic Services PSC Inc., dba The Urology Group, Cincinnati, Ohio
  - University Hospital Case Medical Center, Cleveland, Ohio
  - Institute of Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Urologic Consultants of Southern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Mount Nittany Medical Center Health Services, Inc. dba Mount Nittany Physician Group, State College, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Virginia Women's Center, Richmond, Virginia
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington
  - The Polyclinic, Seattle, Washington

REFERENCES:
- [Derived] McCammon K, Gousse A, Kohan A, Glazier D, Gruenenfelder J, Bai Z, Patel A, Hale D. Early and Consistent Improvements in Urinary Symptoms and Quality of Life With OnabotulinumtoxinA in Patients With Overactive Bladder and Urinary Incontinence: Results From a Randomized, Placebo-controlled, Phase IV Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Jul 1;27(7):450-456. doi: 10.1097/SPV.0000000000000914. PMID 32665528

RESULTS

PARTICIPANT FLOW:
Period: Cycle 1
Arm/Group | OnabotulinumtoxinA | Placebo/OnabotulinumtoxinA
Started | 129 | 125
Completed | 116 | 121
Not Completed | 13 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Personal Reasons | 4 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Other Miscellaneous Reasons | 3 | 1
Period: Cycle 2
Arm/Group | OnabotulinumtoxinA | Placebo/OnabotulinumtoxinA
Started | 88 (Not all participants participated in Cycle 2.) | 107
Completed | 87 | 106
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA | Placebo/OnabotulinumtoxinA | Total
Number analyzed (Participants) | 129 | 125 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (12.73) | 60.9 (12.10) | 60.8 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 112 | 226
  Male | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a 100% Reduction in Urinary Incontinence Episodes
Description: Urinary incontinence is defined as involuntary loss of urine as recorded by the participant in a bladder diary during the 3 consecutive days prior to the study visit in Treatment Cycle 1. The number of incontinence episodes were averaged daily during this period and compared to baseline to determine 100% reduction in episodes.
Time Frame: Baseline, Week 12
Population: Participants from the Intent-to-Treat Population, all participants who were randomized to study drug, with data available at Baseline and Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | OnabotulinumtoxinA | Placebo/OnabotulinumtoxinA
Number analyzed (Participants) | 128 | 125
percentage of participants | 32.0 | 7.2

2. Primary Outcome: Change From Baseline in the Daily Average Number of Episodes of Urinary Incontinence
Description: Urinary incontinence is defined as involuntary loss of urine as recorded by the participant in a bladder diary during the 3 consecutive days prior to the study visit in Treatment Cycle 1. The number of incontinence episodes were averaged daily during this period. A negative number change from Baseline indicates an improvement and a positive number change from Baseline indicates a worsening.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: incontinence episodes
Arm/Group | OnabotulinumtoxinA | Placebo/OnabotulinumtoxinA
Number analyzed (Participants) | 128 | 125
incontinence episodes
  Baseline | 5.4 (3.16) | 5.9 (3.75)
  Change at Week 12 | -3.4 (3.69) | -1.7 (3.23)

3. Secondary Outcome: Change From Baseline in King's Health Questionnaire (KHQ) Domain Scores
Description: The King's Health Questionnaire is a disease-specific questionnaire that measures the quality of life of participants with urinary incontinence. The questionnaire consists of 7 domains, including emotions, personal relationships, physical limitations, role limitations, severity (coping) measures, sleep/energy and social limitations. Domain scores range from 0 to 100, with a lower score indicating a preferable health status (absence of urinary incontinence impacts). A negative number change from Baseline indicates improvement and a positive number change from Baseline indicates a worsening.
Time Frame: Baseline, Week 12
Population: Intent-to-Treat Population included all participants who were randomized to study drug, "n" is the number of participants with available data at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OnabotulinumtoxinA | Placebo/OnabotulinumtoxinA
Number analyzed (Participants) | 129 | 125
score on a scale
  Emotions, Baseline (n=128,123) | 52.38 (30.982) | 53.60 (29.243)
  Emotions, Change at Week 12 (n=121,118) | -21.98 (33.164) | -6.63 (26.177)
  Personal Relationships, Baseline (n=87,86) | 42.91 (35.000) | 43.22 (36.638)
  Personal Relationships,Change at Week 12 (n=71,74) | -18.31 (31.390) | -6.98 (28.537)
  Physical Limitations, Baseline (n=128,125) | 66.41 (29.651) | 64.93 (30.145)
  Physical Limitations,Change at Week 12 (n=121,120) | -32.37 (35.046) | -10.00 (28.039)
  Role Limitations, Baseline (n=127,123) | 70.73 (27.516) | 71.95 (29.362)
  Role Limitations, Change at Week 12 (n=117,117) | -37.75 (32.928) | -16.67 (28.196)
  Severity (Coping) Measures, Baseline (n=128,124) | 65.68 (21.347) | 69.18 (22.201)
  Severity (Coping), Change at Week 12 (n=121,119) | -24.89 (29.558) | -9.17 (19.925)
  Sleep/Energy, Baseline (n=128,123) | 71.35 (25.696) | 71.00 (25.053)
  Sleep/Energy, Change at Week 12 (n=121,118) | -24.93 (26.885) | -10.03 (25.796)
  Social Limitations, Baseline (n=128,125) | 43.69 (28.911) | 46.81 (32.065)
  Social Limitations, Change at Week 12 (n=120,120) | -20.40 (32.634) | -5.97 (25.332)

4. Secondary Outcome: Change From Baseline in the Daily Average Number of Micturition Episodes
Description: The number of micturition episodes (the number of times a patient urinates into the toilet) in Treatment Cycle 1 was recorded by the participant in a bladder diary during the 3 consecutive days prior to the study visit in Treatment Cycle 1. The number of micturition episodes were averaged daily during this period A negative number change from Baseline indicates an improvement and a positive number change from Baseline indicates a worsening.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micturition episodes
Arm/Group | OnabotulinumtoxinA | Placebo/OnabotulinumtoxinA
Number analyzed (Participants) | 128 | 125
micturition episodes
  Baseline | 10.2 (2.99) | 11.1 (3.43)
  Change at Week 12 | -2.6 (2.71) | -1.3 (2.62)

5. Secondary Outcome: Change From Baseline in the Daily Average Number of Urgency Episodes
Description: The number of daily urgency episodes (the number of times a patient experiences the urgency to urinate) in Treatment Cycle 1 was recorded by the patient in a bladder diary during the 3 consecutive days prior to the study visit in Treatment Cycle 1. The number of urgency episodes were averaged daily during this period A negative number change from Baseline indicates an improvement and a positive number change from Baseline indicates a worsening.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: urgency episodes
Arm/Group | OnabotulinumtoxinA | Placebo/OnabotulinumtoxinA
Number analyzed (Participants) | 128 | 125
urgency episodes
  Baseline | 4.9 (3.09) | 5.3 (3.47)
  Change at Week 12 | -3.3 (3.49) | -1.7 (3.24)

6. Secondary Outcome: Change From Baseline in the Daily Average Number of Nocturia Episodes
Description: Nocturia episodes were recorded by the participant in a bladder diary during the 3 consecutive days prior to the study visit in Treatment Cycle 1. The number of nocturia episodes were averaged daily during this period. A nocturia episode is a void (urinating into the toilet) that interrupts one's sleep. A negative number change from Baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nocturia episodes
Arm/Group | OnabotulinumtoxinA | Placebo/OnabotulinumtoxinA
Number analyzed (Participants) | 128 | 125
nocturia episodes
  Baseline | 2.2 (1.43) | 2.1 (1.43)
  Change at Week 12 | -0.7 (1.34) | -0.4 (1.28)

ADVERSE EVENTS:
Description: The Safety Population, all participants who received at least one dose of study drug, was used to determine the number of participants at risk for Serious Adverse Events and Adverse Events.
Groups:
- OnabotulinumtoxinA (Cycle 1): OnabotulinumtoxinA (BOTOX®) 100 U injected into the detrusor at Day 1 in Cycle 1.
- Placebo (Cycle 1): Placebo (Normal saline) injected into the detrusor on Day 1 of Cycle 1.
- OnabotulinumtoxinA (Cycle 2): OnabotulinumtoxinA (BOTOX®) 100 U injected into the detrusor at Day 1 in Cycle 2.
Arm/Group | OnabotulinumtoxinA (Cycle 1) | Placebo (Cycle 1) | OnabotulinumtoxinA (Cycle 2)
Serious Adverse Events (participants affected / at risk) | 6/128 | 8/125 | 3/195
Other Adverse Events (participants affected / at risk) | 51/128 | 34/125 | 75/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA (Cycle 1) (N=128) | Placebo (Cycle 1) (N=125) | OnabotulinumtoxinA (Cycle 2) (N=195)
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Hernia obstructive (General disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA (Cycle 1) (N=128) | Placebo (Cycle 1) (N=125) | OnabotulinumtoxinA (Cycle 2) (N=195)
Constipation (Gastrointestinal disorders) | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 3 | 0
Oedema peripheral (General disorders) | 0 | 1 | 3
Pyrexia (General disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 27 | 8 | 43
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 3
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 4 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 3 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Residual urine volume increased (Investigations) | 3 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Convulsion (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 8 | 0 | 17
Dysuria (Renal and urinary disorders) | 6 | 3 | 6
Bladder discomfort (Renal and urinary disorders) | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 2
Urethral pain (Renal and urinary disorders) | 2 | 0 | 0
Urinary straining (Renal and urinary disorders) | 2 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.